CLINICAL TRIAL: NCT01831401
Title: A Randomised Controlled Study Investigating the Effect of Patient Pelvic Positioning and Method of Acetabular Component Insertion on Acetabular Component Inclination During Total Hip Arthroplasty (THA).
Brief Title: A Study Investigating the Effect of Patient Pelvic Positioning and Method of Acetabular Component Insertion on Acetabular Component Inclination During Total Hip Arthroplasty (THA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Musgrave Park Hospital (Other)
Collaborators: Belfast Arthroplasty Research Trust (BART) (Unknown); Belfast Health and Social Care Trust (Other); Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Professor David Beverland, Consultant Orthopaedic Surgeon, Musgrave Park Hospital
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 12080DB-SW
Record Dates: First submitted 2013-02-15; First posted 2013-04-15 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Total Hip Arthroplasty; Total Hip Replacement; THA; THR
Keywords: Acetabular component inclination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 0° Head Down (horizontal) & Standard Introducer. (Experimental): Operating table position 0° head down (horizontal) & standard straight acetabular component introducer without alignment guide.
  Interventions: Procedure: Operating table position 0° head down (Horizontal); Device: Standard straight acetabular component introducer without alignment guide.
- 0° Head Down (horizontal) & Modified 35° Introducer. (Experimental): Operating table position 0°head down (horizontal) & modified 35° acetabular component introducer.
  Interventions: Procedure: Operating table position 0° head down (Horizontal); Device: Modified 35° acetabular component introducer.
- 0°Head Down (horizontal) & Inclinometer-assisted Introducer. (Experimental): Operating table position 0°head down (horizontal) & standard straight acetabular component introducer without alignment guide.
  Interventions: Procedure: Operating table position 0° head down (Horizontal); Device: Inclinometer-assisted acetabular component introducer.
- 7° Head Down & Standard Introducer. (Experimental): Operating table position 7° head down & standard straight acetabular component introducer without alignment guide.
  Interventions: Procedure: Operating table position 7° head down.; Device: Standard straight acetabular component introducer without alignment guide.
- 7° Head Down & Modified 35° Introducer. (Experimental): Operating table position 7° head down & modified 35° acetabular component introducer.
  Interventions: Procedure: Operating table position 7° head down.; Device: Modified 35° acetabular component introducer.
- 7° Head Down & Inclinometer-assisted Introducer. (Experimental): Operating table position 7° head down & inclinometer-assisted acetabular component introducer.
  Interventions: Procedure: Operating table position 7° head down.; Device: Inclinometer-assisted acetabular component introducer.
- Y° Head Down & Standard Introducer. (Experimental): Operating table position Y° head down (angle required to obtain vertical Transverse Pelvis Lines) & standard straight acetabular component introducer without alignment guide.
  Interventions: Procedure: Operating table position Y° head down; Device: Standard straight acetabular component introducer without alignment guide.
- Y° Head Down & Modified 35° Introducer. (Experimental): Operating table position Y° head down (angle required to obtain vertical Transverse Pelvis Lines) & modified 35°acetabular component introducer.
  Interventions: Procedure: Operating table position Y° head down; Device: Modified 35° acetabular component introducer.
- Y° Head Down & Inclinometer-assisted Introducer. (Experimental): Operating table position Y° head down (angle required to obtain vertical Transverse Pelvis Lines) & inclinometer-assisted acetabular component introducer.
  Interventions: Procedure: Operating table position Y° head down; Device: Inclinometer-assisted acetabular component introducer.

INTERVENTIONS:
Procedure: Operating table position 0° head down (Horizontal)
  Arms: 0° Head Down (horizontal) & Modified 35° Introducer.; 0° Head Down (horizontal) & Standard Introducer.; 0°Head Down (horizontal) & Inclinometer-assisted Introducer.
Procedure: Operating table position 7° head down.
  Arms: 7° Head Down & Inclinometer-assisted Introducer.; 7° Head Down & Modified 35° Introducer.; 7° Head Down & Standard Introducer.
Procedure: Operating table position Y° head down — Operating table position Y° head down (angle required to obtain vertical Transverse Pelvis Lines).
  Arms: Y° Head Down & Inclinometer-assisted Introducer.; Y° Head Down & Modified 35° Introducer.; Y° Head Down & Standard Introducer.
Device: Standard straight acetabular component introducer without alignment guide.
  Arms: 0° Head Down (horizontal) & Standard Introducer.; 7° Head Down & Standard Introducer.; Y° Head Down & Standard Introducer.
Device: Modified 35° acetabular component introducer.
  Arms: 0° Head Down (horizontal) & Modified 35° Introducer.; 7° Head Down & Modified 35° Introducer.; Y° Head Down & Modified 35° Introducer.
Device: Inclinometer-assisted acetabular component introducer.
  Arms: 0°Head Down (horizontal) & Inclinometer-assisted Introducer.; 7° Head Down & Inclinometer-assisted Introducer.; Y° Head Down & Inclinometer-assisted Introducer.

SUMMARY:
Total Hip Arthroplasty (THA) is one of the most commonly performed orthopaedic operations worldwide. The main aim is overall improvement in levels of patient pain and mobility. Such surgery involves implantation of both an acetabular and femoral component. With the patient in the lateral decubitus position, the Orthopaedic Surgeon assumes that the pelvis is in a neutral position with respect to all three body planes at the time of acetabular component implantation.

With regard to THA, the current orthopaedic literature demonstrates a clear relationship between acetabular component positioning, polyethylene wear and risk of dislocation. Problems with edge loading, stripe wear and squeaking are also associated with higher acetabular inclination angles, particularly in hard-on-hard bearing implants.

The important parameters of acetabular component positioning are depth, height, version and inclination.

Control of acetabular component inclination, particularly in the lateral decubitus position, is difficult and remains a challenge for the Orthopaedic Surgeon.

Accurate implantation of the acetabular component within the 'safe zone' of radiological inclination is dependent on:

* Operative version
* Operative inclination
* Pelvic position (Primarily, but not exclusively, abduction / adduction.)

This study aims to investigate the effect of patient pelvic positioning and method of acetabular component insertion on acetabular component inclination during Total Hip Arthroplasty (THA).

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 16 and 100 years awaiting primary Total Hip Arthroplasty the care of Professor D Beverland and Mr D Molloy in Musgrave Park Hospital will initially be invited to participate.

Exclusion Criteria:

* Patients unable to provide fully informed consent.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Radiological acetabular component inclination. | Radiological acetabular component inclination will be measured on the routine post-operative pelvic x-ray, usually within 48 hrs from time of surgery.
  The study has two primary aims, each with a different primary outcome.
  The first primary aim is to investigate the effect of adjusting patient pelvic position in the transverse plane by using a head down position of the operating table.
  This is to determine, when aiming for 35° of operative inclination, which operating table position most accurately achieves a target radiological inclination of 42° on the post-operative x-ray:
  1. 0° head down (Horizontal),
  2. 7° head down, or
  3. Y° head down (Angle required to obtain vertical Transverse Pelvic Lines).
Operative Acetabular Component Inclination. | Operative acetabular component inclination will be measured intra-operatively.
  The study has two primary aims, each with a different primary outcome.
  The second primary aim is to determine which of the three methods of acetabular component insertion most accurately allows the Orthopaedic Surgeon to obtain the desired operative inclination of 35° during THA when using a cementless cup:
  1. Standard straight introducer without any alignment guide,
  2. Modified 35° introducer with horizontal alignment guide, or
  3. Digital inclinometer assisted introducer.

SECONDARY OUTCOMES:
Proportion of cases in which the target radiological inclination of 42 +/- 5° is actually obtained. | Radiological acetabular component inclination will be measured on the routine post-operative pelvic x-ray, usually within 48 hrs from time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: David E Beverland, MD FRCS(Orth), Principal Investigator — Musgrave Park Hospital / Belfast Health & Social Care Trust
Locations (1):
- Musgrave Park Hospital, Belfast, County Antrim, United Kingdom

REFERENCES:
- [Background] Hill JC, Gibson DP, Pagoti R, Beverland DE. Photographic measurement of the inclination of the acetabular component in total hip replacement using the posterior approach. J Bone Joint Surg Br. 2010 Sep;92(9):1209-14. doi: 10.1302/0301-620X.92B9.24476. PMID 20798436
- [Derived] O'Neill CKJ, Magill P, Hill JC, Patterson CC, Molloy DO, Gill HS, Beverland DE. Correction of pelvic adduction during total hip arthroplasty reduces variability in radiographic inclination: findings of a randomised controlled trial. Hip Int. 2018 May;28(3):240-245. doi: 10.1177/1120700018777480. PMID 30165765
- [Derived] O'Neill CKJ, Hill JC, Patterson CC, Molloy DO, Gill HS, Beverland DE. Reducing variability in apparent operative inclination during total hip arthroplasty: findings of a randomised controlled trial. Hip Int. 2018 May;28(3):234-239. doi: 10.1177/1120700018777485. PMID 30165761